CLINICAL TRIAL: NCT06239662
Title: Therapeutic Education Groups for Childhood Obesity: a Randomized Controlled Trial
Brief Title: Therapeutic Education Groups for Childhood Obesity
Acronym: GET-Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GET-Obesità N.01-18/02/16
Record Dates: First submitted 2023-12-28; First posted 2024-02-02 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-10

CONDITIONS: Childhood Obesity
Keywords: Childhood obesity; Group Intervention; Psychological Aspects
MeSH Terms: conditions — Pediatric Obesity | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic group intervention (Experimental): Patients will be called in groups every 3 months for a total of 10 meetings. At each meeting they will be weighed and measured. Each meeting will focus on a topic of nutritional/lifestyle interest and will see the co-presence of the figures of the dietician and the psychologist, in order to allow an emotional declination for all the participants.
  Interventions: Behavioral: Therapeutic Group
- Usual care (Active Comparator): Patients will be called individually every 3 months for a total of 10 meetings. At each meeting they will be weighed and measured. Each meeting will focus on a topic of nutritional/lifestyle interest. The meetings will be conducted by a dietician.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Therapeutic Group — The first part of each meeting, lasting 45 minutes, will be held only with children and young people, while parents will wait in the waiting room. At the end of the first part, for each meeting, the children will be asked to make a commitment relating to the topics covered, which will be verified in the following meeting. Once the part with the patients has concluded, they will be accompanied to an adjacent environment where a pediatrician volunteer will be waiting for them and will offer fun and socialization activities. In the meantime, the parents will be seated and will address, together with the team staff, the same issues discussed with their children, again for a duration of approximately 45 minutes. Parents will also be invited to make a commitment similar to that required of children.
  Arms: Therapeutic group intervention
Behavioral: Usual care — The dietician will meet individually each child together with parents. Dietician will provide nutritional advices.
  Arms: Usual care

SUMMARY:
The goal of this clinical trial is to test the efficacy of an educational therapeutic intervention in treating obesity in a pediatric population.

It aims to verify the differences between the experimental group (group-based program) and the control group (individual program) in respect to the BMI z-score values between baseline measurement (beginning of treatment), final measurement (end of treatment) and 18 months follow-up.

DETAILED DESCRIPTION:
One of the aim of this clinical trial is to verify that the direct management of the emotional and relational aspects of patients and family plays an important role in maintaining the weight changes achieved in the long term.

The potential added value of the present study concerns the better understanding of the role of psychological and emotional aspects in the treatment of childhood obesity and in maintaining results in the long term.

The clinical trial aims to recruit 300 obese children randomized in two groups: experimental group and control group.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (>= 95th percentile);
* No organic causes of obesity;
* Sufficient understanding and production of Italian language;
* Age between 7 and 17 years old;
* Absence of neuropsychiatric diagnosis;
* Subscription of the Informed Consent from both parents (or legal guardian).

Exclusion Criteria

* Degree of obesity< 95th percentile;
* Organic causes of obesity;
* Insufficient understanding and production of Italian language;
* Age <7 or >17;
* Presence of neuropsychiatric diagnosis;
* One parent (or legal guardian) refuses to subscribe the Informed Consent.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
BMI z-score | measurement at end of treatment i.e approximately 24 months after baseline measurements
  BMI z-score variation from baseline to end of treatment
BMI z-score | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  BMI z-score variation from baseline to 18 months after the and of treatment

SECONDARY OUTCOMES:
healthy dietary habits | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in the daily consumption (in frequency) of fruits and vegetables measurement at end of treatment i.e approximately 24 months after baseline measurements
healthy dietary habits | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in the daily consumption (in frequency) of fruits and vegetables measurement from baseline to 18 months after the and of treatment
unhealthy dietary habits | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in the weekly consumption (in frequency) of packed and high-calorie food measurment at end of treatment i.e approximately 24 months after baseline measurements
unhealthy dietary habits | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in the weekly consumption (in frequency) of packed and high-calorie food measurment from baseline to 18 months after the and of treatment
Biohumoral exams from blood sample: Uric acid | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in the value measurements (differences expressed in mg/dL) at end of treatment i.e approximately 24 months after baseline measurements
Biohumoral exams from blood sample: Transaminases | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in the value measurements (differences expressed in U/l) at end of treatment i.e approximately 24 months after baseline measurements
Biohumoral exams from blood sample: Glycemia | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in the value measurements (differences expressed in mg/dL) at end of treatment i.e approximately 24 months after baseline measurements
Biohumoral exams from blood sample: Insulin | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in the value measurements (differences expressed in µU/mL) at end of treatment i.e approximately 24 months after baseline measurements
Biohumoral exams from blood sample: Glycated hemoglobin | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in the value measurements (differences expressed mmol/moli) at end of treatment i.e approximately 24 months after baseline measurements
Biohumoral exams from blood sample: Cholesterol | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in the value measurements (differences expressed mg/dL) at end of treatment i.e approximately 24 months after baseline measurements
Biohumoral exams from blood sample: Triglycerides | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in the value measurements (differences expressed mg/dL) at end of treatment i.e approximately 24 months after baseline measurements
Biohumoral exams from blood sample: Thyroid-stimulating hormone | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in the value measurements (differences expressed μIU/ml) at end of treatment i.e approximately 24 months after baseline measurements
Biohumoral exams from blood sample: Uric acid | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in the value measurements (differences expressed in mg/dL) from baseline to 18 months after the and of treatment
Biohumoral exams from blood sample: Transaminases | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in the value measurements (differences expressed in U/l) from baseline to 18 months after the and of treatment
Biohumoral exams from blood sample: Glycemia | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in the value measurements (differences expressed in mg/dL) from baseline to 18 months after the and of treatment
Biohumoral exams from blood sample: Insulin | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in the value measurements (differences expressed in µU/mL) from baseline to 18 months after the and of treatment
Biohumoral exams from blood sample: Glycated hemoglobin | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in the value measurements (differences expressed in mmol/moli) from baseline to 18 months after the and of treatment
Biohumoral exams from blood sample: Cholesterol | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in the value measurements (differences expressed in mg/dL) from baseline to 18 months after the and of treatment
Biohumoral exams from blood sample: Triglycerides | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in the value measurements (differences expressed in mg/dL) from baseline to 18 months after the and of treatment
Biohumoral exams from blood sample: Thyroid-stimulating hormone | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in the value measurements (differences expressed in μIU/ml) from baseline to 18 months after the and of treatment
Psychological questionnaire TAS-20 (Toronto Alexithymia Scale) | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in TAS-20 overall and sub-scale scores (differences) from baseline to the end of treatment i.e approximately 24 months after baseline measurements.Scoring range: 20-100; cutoff 60 (higher scores indicate greater impairment/challenges).
Psychological questionnaire TAS-20 (Toronto Alexithymia Scale) | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in TAS-20 overall and sub-scale scores (differences) from baseline to approximately 18 months after the end of treatment. Scoring range: 20-100; cutoff 60 (higher scores indicate greater impairment/challenges).
Psychological questionnaire PEDSQL (Pediatric Quality of life) | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in PEDSQL overall and sub-scale scores (differences) from baseline to the end of treatment i.e approximately 24 months after baseline measurements. Scores are linearly transformed to a 0-100 scale in which high score means better condition.
Psychological questionnaire PEDSQL (Pediatric Quality of life) | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in PEDSQL overall and sub-scale scores (differences) from baseline to approximately 18 months after the end of treatment. Scores are linearly transformed to a 0-100 scale in which high score means better condition.
Psychological questionnaire CBCL (Child Behaviour Checklist) | measurement at end of treatment i.e approximately 24 months after baseline measurements
  variation in CBCL overall and sub-scale scores (differences) from baseline to the end of treatment i.e approximately 24 months after baseline measurements. Scores below the 93rd percentile is considered normal, scores between the 93-97th percentile are borderline clinical, and scores above the 97th percentile are in the clinical range.
Psychological questionnaire CBCL (Child Behaviour Checklist) | measurement at 18 months after the end of treatment i.e approximately 42 months after baseline measurements
  variation in CBCL overall and sub-scale scores (differences) from baseline to approximately 18 months after the end of treatment. Scores below the 93rd percentile is considered normal, scores between the 93-97th percentile are borderline clinical, and scores above the 97th percentile are in the clinical range
Drop-out | measurement at end of treatment i.e approximately 24 months after baseline measurements
  qualitative differences between experimental and control group in drop-out per cent

CONTACTS AND LOCATIONS:
Overall Officials: Marta Fontana, Psycologist, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia

IPD SHARING:
Plan to Share IPD: Undecided
We do not have the authorization to share IPD. We are in the process to agree with the Ethic Committee how the share data.

REFERENCES:
- [Background] Panebianco D, Gallupe O, Carrington PJ, Colozzi I. Personal support networks, social capital, and risk of relapse among individuals treated for substance use issues. Int J Drug Policy. 2016 Jan;27:146-53. doi: 10.1016/j.drugpo.2015.09.009. Epub 2015 Sep 28. PMID 26520237
- [Background] Kalavainen MP, Korppi MO, Nuutinen OM. Clinical efficacy of group-based treatment for childhood obesity compared with routinely given individual counseling. Int J Obes (Lond). 2007 Oct;31(10):1500-8. doi: 10.1038/sj.ijo.0803628. Epub 2007 Apr 17. PMID 17438555
- [Background] Zeller M, Daniels S. The obesity epidemic: family matters. J Pediatr. 2004 Jul;145(1):3-4. doi: 10.1016/j.jpeds.2004.04.038. No abstract available. PMID 15238894
- [Background] Braet C, Mervielde I, Vandereycken W. Psychological aspects of childhood obesity: a controlled study in a clinical and nonclinical sample. J Pediatr Psychol. 1997 Feb;22(1):59-71. doi: 10.1093/jpepsy/22.1.59. PMID 9019048
- [Background] French SA, Story M, Jeffery RW. Environmental influences on eating and physical activity. Annu Rev Public Health. 2001;22:309-35. doi: 10.1146/annurev.publhealth.22.1.309. PMID 11274524
- [Background] Trombini E, Baldaro B, Bertaccini R, Mattei C, Montebarocci O, Rossi N. Maternal attitudes and attachment styles in mothers of obese children. Percept Mot Skills. 2003 Oct;97(2):613-20. doi: 10.2466/pms.2003.97.2.613. PMID 14620250
- [Background] Goldfield GS, Mallory R, Parker T, Cunningham T, Legg C, Lumb A, Parker K, Prud'homme D, Adamo KB. Effects of modifying physical activity and sedentary behavior on psychosocial adjustment in overweight/obese children. J Pediatr Psychol. 2007 Aug;32(7):783-93. doi: 10.1093/jpepsy/jsm017. Epub 2007 Apr 19. PMID 17449466
- [Background] Braet C, Tanghe A, Decaluwe V, Moens E, Rosseel Y. Inpatient treatment for children with obesity: weight loss, psychological well-being, and eating behavior. J Pediatr Psychol. 2004 Oct;29(7):519-29. doi: 10.1093/jpepsy/jsh054. PMID 15347700
- [Background] Hingle MD, O'Connor TM, Dave JM, Baranowski T. Parental involvement in interventions to improve child dietary intake: a systematic review. Prev Med. 2010 Aug;51(2):103-11. doi: 10.1016/j.ypmed.2010.04.014. Epub 2010 May 10. PMID 20462509
- [Background] Fonseca H, Palmeira AL, Martins SC, Falcato L, Quaresma A. Managing paediatric obesity: a multidisciplinary intervention including peers in the therapeutic process. BMC Pediatr. 2014 Apr 3;14:89. doi: 10.1186/1471-2431-14-89. PMID 24693926
- [Background] Kader M, Sundblom E, Elinder LS. Effectiveness of universal parental support interventions addressing children's dietary habits, physical activity and bodyweight: A systematic review. Prev Med. 2015 Aug;77:52-67. doi: 10.1016/j.ypmed.2015.05.005. Epub 2015 May 14. PMID 25981555
- [Background] Wilfley DE, Tibbs TL, Van Buren DJ, Reach KP, Walker MS, Epstein LH. Lifestyle interventions in the treatment of childhood overweight: a meta-analytic review of randomized controlled trials. Health Psychol. 2007 Sep;26(5):521-32. doi: 10.1037/0278-6133.26.5.521. PMID 17845100
- [Background] Epstein LH, Leddy JJ, Temple JL, Faith MS. Food reinforcement and eating: a multilevel analysis. Psychol Bull. 2007 Sep;133(5):884-906. doi: 10.1037/0033-2909.133.5.884. PMID 17723034
- [Background] Davoli AM, Broccoli S, Bonvicini L, Fabbri A, Ferrari E, D'Angelo S, Di Buono A, Montagna G, Panza C, Pinotti M, Romani G, Storani S, Tamelli M, Candela S, Giorgi Rossi P. Pediatrician-led motivational interviewing to treat overweight children: an RCT. Pediatrics. 2013 Nov;132(5):e1236-46. doi: 10.1542/peds.2013-1738. Epub 2013 Oct 21. PMID 24144717
- See also: BMI definition — https://www.cdc.gov/index.htm
- See also: national surveillance system Okkio alla SALUTE — https://www.cdc.gov/index.htm